CLINICAL TRIAL: NCT00185198
Title: Multicenter, Double Blind, Randomized, Placebo Controlled Study of Testogel® (Testosterone 50-100mg) to Evaluate Its Efficacy and Safety in Men Presenting With Typical Symptoms of Partial Androgen Deficiency of Aging Males (PADAM) Over a Period of 6 Months With 12 Months Open Label Follow-up
Brief Title: Efficacy and Safety of Testogel® in Men With Partial Androgen Deficiency of Aging Males (PADAM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91297; 2004-001545-15 (EudraCT Number); 307720 (Other: Company internal)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Androgens (Deficiency); Male
Keywords: Partial androgen deficiency of aging males (PADAM)
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Testogel (Testosterone, BAYV001915)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testogel (Testosterone, BAYV001915) — 50mg (5g gel sachet), 75mg (5g+2.5g sachet) or 100mg (2x5g sachet) per day applied to the skin of the shoulders, arms or abdomen for 18 months
  Arms: Arm 1
Drug: Placebo — 5g gel sachet, 5g+2.5g sachet or 2x5g sachets per day applied to the skin of the shoulders, arms or abdomen for 6 months followed by 12 months treatment with testosterone 1% gel as described for arm 1
  Arms: Arm 2

SUMMARY:
The purpose of this study is to investigate the effect of a testosterone replacement therapy called Testogel in men with PADAM. The effects on body composition (lean, fat and bone) and other symptoms of PADAM and safety will be studied.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic hypogonadism
* Willing to avoid significant change in the pattern of physical exercise and lifestyle for the duration of the study

Exclusion Criteria:

* Patients with any contraindication for testosterone use

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Lean body mass at 6 months | baseline, month 6 and month 18

SECONDARY OUTCOMES:
Change in total body mass, fat mass and bone density | baseline, month 6 and month 18
Evaluation of symptoms by the aging males symptoms rating scale | baseline, month 6 and month 18
Change in testosterone | baseline, month 6 and month 18
Safety parameters | baseline, month 6 and month 18

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Austria (5):
  - Vienna, Vienna
  - Graz
  - Innsbruck
  - Salzburg
  - Vienna
- Finland (3):
  - Helsinki
  - Oulu
  - Tampere
- Germany (5):
  - Bonn, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg
- Dublin, Ireland
- Italy (3):
  - Milan
  - Napoli
  - Roma
- Spain (3):
  - L'Hospitalet de Llobregat, Barcelona
  - Madrid, Madrid
  - Barcelona
- Sweden (3):
  - Gothenburg
  - Malmo
  - Stockholm
- United Kingdom (5):
  - Reading, Berkshire
  - Wigan, Manchester
  - Cardiff
  - London
  - Sheffield